CLINICAL TRIAL: NCT04821271
Title: An Investigation of the Antidepressant Effects of the mGlu2/3 Receptor Antagonist TS-161 in Treatment-Resistant Depression
Brief Title: Antidepressant Effects of TS-161 in Treatment-Resistant Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to low recruitment
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10000101; 000101-M
Record Dates: First submitted 2021-02-27; First posted 2021-03-29 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder; Treatment-Resistant Depression; Depression
Keywords: Biomarker; Neurobiology; Glutamate; Magnetoencephalography; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TS-161, then Placebo (Experimental): Participants with major depressive disorder (MDD) were randomized to receive TS-161 100mg capsule orally once per day for three weeks (with option to decrease to 50 mg due to drug intolerance), followed by Placebo capsule orally once per day for three weeks.
  Interventions: Other: Placebo; Drug: TS-161
- Placebo, then TS-161 (Experimental): Participants with major depressive disorder (MDD) were randomized to receive Placebo capsule orally once per day for three weeks, followed by TS-161 100mg capsule orally once per day for three weeks (with option to decrease to 50 mg due to drug intolerance).
  Interventions: Other: Placebo; Drug: TS-161

INTERVENTIONS:
Other: Placebo — Participants received Placebo capsule orally once daily for three weeks.
Drug: TS-161 — Participants received TS-161 50-100 mg capsule orally once daily for three weeks. TS-161 is a mGlu2/3 receptor antagonist prodrug.

SUMMARY:
Background:

Major depressive disorder (MDD) is a common, chronic mental illness. It can take weeks to months for antidepressants to work. Researchers want to test a new drug that might act more rapidly.

Objective:

To see if TS-161 will improve symptoms of depression in people with MDD.

Eligibility:

Adults ages 18-65 with MDD without psychotic features.

Design:

Participants will be screened under a separate protocol. They will have blood tests. They will complete surveys about their symptoms.

Participants will have an inpatient visit at NIH. Participation may last 12-16 weeks.

During the first phase of the study, participants will be tapered off their psychiatric medicines. For 2 weeks they will have a drug-free period.

During Phase II participants will take TS-161 or placebo. They will take TS-161 for 3 weeks and placebo for 3 weeks. In between the 3-week time period, they will have 2-3 weeks where they will be drug free. Participants will also have the following tests during this time:

* Interviews
* Physical exams
* Psychological tests and surveys about their symptoms
* Blood draws and urine samples
* They may complete tests of mood and thinking
* Magnetic resonance imaging (MRI): Participants will lie in a machine that takes pictures of their brain.
* Functional MRIs: They will perform tasks displayed on a computer screen inside the MRI scanner
* Magnetoencephalography (MEG): Participants will lie down and do tasks of memory, attention, and thinking. A cone lowered on their head will record brain activity.
* Electrocardiograms to record the heart s electrical activity. Electrodes will be placed on the skin....

DETAILED DESCRIPTION:
OBJECTIVE

Modulation of glutamatergic signaling is implicated in improvement of depressive symptoms and related constructs/dimensions of observable behavior and neurobiological measures with treatment. Current standard monoaminergic pharmacological approaches for major depressive disorder (MDD) have proven to be only modestly effective during acute major depressive episodes (MDEs). We have systematically tested different glutamatergic modulators in subjects with mood disorders in order to develop improved therapeutics. We found that the N-methyl-D-aspartate receptor (NMDAR) antagonist, ketamine, produces rapid antidepressant effects in patients with treatment-resistant depression (TRD in MDD, Bipolar Disorder) and in suicidal ideation. However, despite being highly efficacious, ketamine produces psychotomimetic effects and has the risk of abuse. The antidepressant effects of mGlu2/3 receptor antagonists are worthy of pursuit, since the antidepressant profile in preclinical assays as well as the synaptic/neural cellular and molecular mechanisms involved in their actions are comparable to those of ketamine, but without the side effects and abuse potential of ketamine.

In the present protocol, we aim to evaluate a new glutamate-mediated mechanism associated with antidepressant efficacy by targeting the mGlu2/3 receptor with a potent and selective antagonist. Targeting the mGlu2/3 receptor with an antagonist is anticipated to, and similar to ketamine, result via pre-synaptic mechanisms in a "glutamate surge" with subsequent alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) activation and gamma power increases but without potential adverse effects that occur with ketamine.

The present Phase 2 proof-of-concept (POC) study is designed to evaluate in subjects with MDD, the antidepressant effects of TS-161, the prodrug of a potent and selective mGlu2/3 receptor antagonist TP0178894 that crosses the blood brain barrier (BBB). In animal model assays of antidepressant efficacy, TS-161 induced acute and prolonged antidepressant-like effects without exhibiting ketamine-like side effects as determined by the lack of increase in locomotor activity or abuse potential.

We will also evaluate the putative neurobiological mechanisms involved in the antidepressant response to TS-161. We expect that this effect may modulate glutamate transmission and reverse the clinical symptoms of depression. The demonstration that an mGlu2/3 receptor antagonist produces antidepressant effects without psychotomimetic side effects would support the therapeutic relevance of the mGlu2/3 receptor and could direct the development of novel drug targets for the treatment of depression.

STUDY POPULATION

Twenty-five individuals with treatment-resistant major depressive disorder (MDD) will be consented.

DESIGN

Male and female subjects, ages 18 to 65 years, with a diagnosis of MDD, currently in an episode of major depression, will be recruited for this study. This study will consist of a randomized, double-blind crossover administration of either the mGlu2/3 receptor antagonist prodrug TS-161 (50 to 100 mg/day given orally) or placebo for 3 weeks. The study will assess the efficacy in improving overall depressive symptomatology and tolerability of TS-161 in treatment-resistant MDD. Other aims of the study include determining whether changes in gamma power obtained via magnetoencephalography (MEG), brain neurochemicals (e.g. glutamate) obtained via magnetic resonance spectroscopy (MRS), and peripheral measures correlate with drug effects and/or antidepressant response to TS-161 in subjects with treatment-resistant MDD.

OUTCOME MEASURES

Primary: Montgomery-Asberg Depression Rating Scale (MADRS) total score.

Secondary: Proportion of subjects achieving remission (MADRS<=10) and response (>=50% reduction from baseline in MADRS total score); change from baseline on the Hamilton Rating Scale (HDRS), change from baseline in Hamilton Anxiety Rating Scale (HAM-A), and the Columbia Suicide Severity Rating Scale (C-SSRS) total scores. Surrogate biomarkers of drug effect/response include: changes in gamma power measured with MEG, changes in prefrontal glutamate levels measured with 7T 1H-MRS, resting and task based functional connectivity with fMRI, neurocognitive functioning, and changes in peripheral biological indices (neurotrophic factors, cell cycle/signal transduction regulators, neuroinflammatory, neuroendocrinological measures, and metabolomic and proteomic measures).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants may be eligible for this study if they:

1. Are able to understand the study and can provide your own consent.
2. Are willing to undergo all study procedures and are available for the duration of the study.
3. Are aged 18 to 65.
4. Have major depressive disorder.
5. Have a current episode of depression lasting at least 4 weeks.
6. Ability to take oral medication.
7. Have not responded to at least one antidepressant.
8. For females of reproductive potential: use of contraception while in the study and for an additional 4 weeks after stopping the study drug.
9. For males of reproductive potential: use of condoms or other types of birth control with partner while in the study and for an additional 3 months after stopping the study drug.
10. Agree to be hospitalized at the NIH Clinical Center.
11. Abstain from alcohol and drug use while in the study.

EXCLUSION CRITERIA:

Participants may not be eligible for this study if they:

1. Are taking any medications that might make it unsafe for you to receive TS-161 or might interfere with our study results.
2. Have been treated with a reversible monoamine oxidase inhibitor (such as phenelzine (Nardil) and tranylcypromine (Parnate)), clozapine, or electroconvulsive therapy (ECT) less than 4 weeks before Phase II.
3. Have been treated with fluoxetine, aripiprazole, or brexpiprazole less than 5 weeks before Phase II.
4. Have ever undergone deep brain stimulation.
5. Have taken ketamine or esketamine for the treatment of depression but did not respond.
6. Are unwilling to stop undergoing one-on-one psychotherapy for the duration of the study.
7. Are pregnant or plan to become pregnant in the next 12 to 16 weeks while in the study, or are breast-feeding.
8. Have schizophrenia or any other psychotic disorder.
9. Had significant drug or alcohol dependence or abuse in the past 3 months (except for nicotine or caffeine), or are currently using illicit substances.
10. Have been diagnosed with borderline or antisocial personality disorder.
11. Had a head injury that caused a loss of consciousness for more than 5 minutes (for the brain imaging).
12. Have a medical illness that might make your participation unsafe, such as heart (including coronary artery disease, atherosclerotic ischemic stroke, and atrial fibrillation), liver, respiratory, blood, immune, or kidney disease or a seizure disorder, based on our evaluation.
13. Have abnormal results on blood and urine tests we will do.
14. Have significant suicidal or homicidal thoughts.
15. Have a positive HIV test.
16. For brain imaging: Have metal in your body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if you were a welder or metal worker, since you may have small metal fragments in the eye.
17. Weigh over 245 lbs. and cannot fit into the MRI scanner.
18. Have a positive, or suspected positive, Coronavirus Disease 2019 (COVID-19) test.
19. Are an National Institute of Mental Health (NIMH) staff member or an immediate family member of an NIMH staff member.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.Clinical and demographic and biomarker participant data collected during the trial, after deidentification.
Supporting Information: SAP
Time Frame: Starting within one year of completion of the study.
Access Criteria: Branch Chief will review requests and access will need to be approved by the NIMH/DIRP SD and OCD NIMH and the NIH Institutional Review Board (IRB).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000101-M.html

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | TS-161, Then Placebo | Placebo, Then TS-161
Started | 6 | 5
TS-161 100mg Then 50mg | 1 | 0
Completed | 4 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Period 2
Arm/Group | TS-161, Then Placebo | Placebo, Then TS-161
Started | 4 | 5
TS-161 100mg, Then 50mg, Then 100mg | 0 | 1
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: Participants with major depressive disorder (MDD) were randomized to receive either TS-161 100mg (with option to dose to 50 mg due to drug intolerance) or Placebo capsule orally once per day for three weeks followed by subsequent intervention for three weeks.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: Change in the Montgomery-Asberg Depression Rating Scale (MADRS) total score from baseline and day 21 (week 3). The MADRS is a 10-item clinician-rated questionnaire to evaluate depressive symptoms in adults and for the assessment of any changes to those symptoms. Each item is rated on a scale of 0 to 6 (0 = absent, 6 = severe) with total score range between 0 and 60. Higher score indicates worsening depression. For each crossover period, the MADRS was completed 60 minutes before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Analysis was the change in total score between baseline and day 21. Change was calculated as the estimated marginal MADRS total score means using a linear mixed model regression.
Time Frame: Baseline and day 21 (week 3)
Population: Analyses based on the intent-to-treat (ITT) population and included all randomized participants who had at least one post-baseline assessment.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- TS-161: Participants with major depressive disorder (MDD) were randomized to receive TS-161 100mg capsule orally once per day for three weeks (with option to decrease to 50 mg due to drug intolerance).
- Placebo: Participants with major depressive disorder (MDD) were randomized to receive Placebo capsule orally once per day for three weeks.
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 28.02 (1.9) | 27.79 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; The null hypothesis was that there would not be treatment differences in mean MADRS total score. Linear mixed model regression using fixed effects of time, treatment, and a time-by-treatment allowed treatment effect estimates to vary by time. The model also included period specific baseline scores, average per person baseline scores (to avoid cross level bias), and period (first or second). All continuous covariates were mean centered. Alpha level of 0.05, and hypothesis was two-sided; Test type: Other — Treatment comparison; p = 0.91, T-test of estimated marginal means

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: Montgomery-Asberg Depression Rating Scale (MADRS) mean total score at 230 minutes and 1, 2, 3, 7, and 14 days following the first treatment administration. The MADRS is a 10-item clinician-rated questionnaire to evaluate depressive symptoms in adults and for the assessment of any changes to those symptoms. Each item is rated on a scale of 0 to 6 (0 = absent, 6 = severe) with total score range between 0 and 60. Higher score indicates worsening depression. For each crossover period, the MADRS was completed 60 minutes before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal means at 230 minutes and 1, 2, 3, 7, and 14 days following the first treatment administration were calculated using a linear mixed model regression.
Time Frame: 230 minutes following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 26.39 (1.82) | 25.01 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.47, T-test of estimated marginal means

3. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: as for outcome 2
Time Frame: Day 1 following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 28.49 (1.82) | 25.68 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.14, T-test of estimated marginal means

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: as for outcome 2
Time Frame: Day 2 following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 28.8 (1.90) | 25.79 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.12, T-test of estimated marginal means

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: as for outcome 2
Time Frame: Day 3 following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 27.91 (1.90) | 27.12 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.69, T-test of estimated marginal means

6. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: as for outcome 2
Time Frame: Day 7 following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 26.59 (1.82) | 27.24 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.73, T-test of estimated marginal means

7. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Mean Total Score
Description: as for outcome 2
Time Frame: Day 14 following the first treatment dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale | 29.13 (1.90) | 27.01 (1.62)
Statistical Analysis 1: Comparison: TS-161 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Treatment comparison; p = 0.28, T-test of estimated marginal means

8. Secondary Outcome: Number of Participants Who Met Remission Criteria at Any Time Point
Description: Number of participants who met remission criteria at any time point after intervention. Remission was defined as Montgomery-Asberg Depression Rating Scale (MADRS) total score ≤10 after intervention. The MADRS is a 10-item clinician-rated questionnaire to evaluate depressive symptoms in adults and for the assessment of any changes to those symptoms. Each item is rated on a scale of 0 to 6 (0 = absent, 6 = severe) with total score range between 0 and 60. Higher score indicates worsening depression. For each crossover period, the MADRS was completed 60 minutes before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose.
Time Frame: Up to three weeks after each intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Met Response Criteria
Description: Number of participants who met response criteria at any timepoint after intervention. Response was defined as a ≥50% reduction from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a 10-item clinician-rated questionnaire to evaluate depressive symptoms in adults and for the assessment of any changes to those symptoms. Each item is rated on a scale of 0 to 6 (0 = absent, 6 = severe) with total score range between 0 and 60. Higher score indicates worsening depression. For each crossover period, the MADRS was completed 60 minutes before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose.
Time Frame: Up to three weeks after each intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

10. Secondary Outcome: Hamilton Depression Rating Scale (HDRS) Mean Total Scores
Description: The Hamilton Depression Rating Scale (HDRS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. HDRS is a widely used observational rating measure of depression severity. The HDRS contains 21 items, but four questions are not added to the numerical total score. The first 17 items are scored on a 3 (0-2) or 5 (0-4) point scale, with total score range between 0 and 52. Scores of 0-7 are considered normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression. For each crossover period, the HDRS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal HDRS total score means were calculated using a linear mixed model regression that controlled for baseline HDRS and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 20.48 (1.71) | 18.21 (1.63)
  Day 1 | 19.78 (1.71) | 18.32 (1.63)
  Day 2 | 20.99 (1.76) | 18.65 (1.63)
  Day 3 | 21.99 (1.76) | 19.88 (1.63)
  Day 7 | 19.58 (1.71) | 19.88 (1.63)
  Day 14 | 22.55 (1.76) | 20.43 (1.63)
  Day 21 | 21.77 (1.76) | 20.76 (1.63)

11. Secondary Outcome: Hamilton Psychiatric Rating Scale for Anxiety (HAM-A) Mean Total Scores
Description: The Hamilton Psychiatric Rating Scale for Anxiety (HAM-A) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. HAM-A is a widely used observational rating measure of anxiety severity. This scale was administered to assess the severity of anxiety and its improvement during the course of therapy. The scale consists of 14 items. Each item is rated on a scale of 0 to 4, with total score range between 0 and 56. A higher score represents greater symptom severity. Total score <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe severity. For each crossover period, the HAM-A was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal HAM-A total score means were calculated using a linear mixed model regression that controlled for baseline HAM-A and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 10.12 (1.16) | 8.73 (1.09)
  Day 1 | 10.32 (1.16) | 10.28 (1.09)
  Day 2 | 11.85 (1.21) | 9.84 (1.09)
  Day 3 | 13.18 (1.21) | 12.62 (1.09)
  Day 7 | 10.02 (1.16) | 12.62 (1.09)
  Day 14 | 11.29 (1.21) | 11.17 (1.09)
  Day 21 | 10.74 (1.21) | 12.73 (1.09)

12. Secondary Outcome: Snaith-Hamilton Pleasure Scale (SHAPS) Mean Total Scores
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. The SHAPS is a 14-item self-report measure of hedonic or pleasurable experiences or the lack of hedonic experiences (e.g., interests, social interactions, or sensory experiences) in adults and for assessment of any changes. Each item is rated on a scale of 1 to 4 (1 = definitely agree or strongly agree, 4 = strongly disagree) with total score range between 14 and 56. Lower scores indicate greater levels of anhedonia. For each crossover period, the SHAPS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal SHAPS total score means were calculated using a linear mixed model regression that controlled for baseline SHAPS and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 36.86 (1.3) | 36.92 (1)
  Day 1 | 36.26 (1.3) | 35.47 (1)
  Day 2 | 37.52 (1.34) | 37.03 (1)
  Day 3 | 39.74 (1.34) | 37.92 (1)
  Day 7 | 38.26 (1.3) | 37.8 (1)
  Day 14 | 39.07 (1.34) | 38.36 (1)
  Day 21 | 39.29 (1.34) | 37.36 (1)

13. Secondary Outcome: Temporal Experience of Pleasure Scale (TEPS) Mean Total Scores
Description: The Temporal Experience of Pleasure Scale (TEPS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. The TEPS is an 18-item self-report measure of consummatory and anticipatory experiences of pleasure or lack of pleasure (i.e., anhedonia) in adults and for the assessment of any changes. Each item is rated on a scale of 0 to 6 (0 = very true for me, 6 = very false for me) with total score range between 0 and 108. Lower scores indicate greater levels of anhedonia. For each crossover period, the TEPS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal TEPS total score means were calculated using a linear mixed model regression that controlled for baseline TEPS and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 48.23 (2.02) | 51.51 (3.16)
  Day 1 | 49.93 (2.03) | 51.29 (2.83)
  Day 2 | 47.6 (1.75) | 49.07 (3.11)
  Day 3 | 46.68 (1.31) | 49.4 (2.65)
  Day 7 | 46.63 (2.34) | 48.07 (3.7)
  Day 14 | 46.51 (2.64) | 48.29 (3.62)
  Day 21 | 46.7 (2.6) | 48.18 (3.65)

14. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Mean Total Score - Positive Affect
Description: The Positive and Negative Affect Schedule (PANAS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. The PANAS is a questionnaire that assesses both positive and negative affect and consists of 20 items, 10 measuring positive affect (e.g., "excited") and 10 measuring negative affect (e.g., "upset"). Each item is rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely) with a total score ranging between 10 and 50 for each affect subscale. Higher scores indicate higher levels of positive or negative affect depending on the subscale. For each crossover period, the PANAS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal total score means were calculated for the positive affect using a linear mixed model regression that controlled for baseline and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 16.91 (1.12) | 18.11 (1.36)
  Day 1 | 18.01 (1.12) | 18.33 (1.36)
  Day 2 | 15.58 (1.16) | 17.77 (1.36)
  Day 3 | 15.58 (1.16) | 16.66 (1.36)
  Day 7 | 15.81 (1.12) | 15.77 (1.36)
  Day 14 | 15.47 (1.16) | 17.77 (1.36)
  Day 21 | 16.91 (1.16) | 17 (1.36)

15. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Mean Total Score - Negative Affect
Description: The Positive and Negative Affect Schedule (PANAS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. The PANAS is a questionnaire that assesses both positive and negative affect and consists of 20 items, 10 measuring positive affect (e.g., "excited") and 10 measuring negative affect (e.g., "upset"). Each item is rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely) with a total score ranging between 10 and 50 for each affect subscale. Higher scores indicate higher levels of positive or negative affect depending on the subscale. For each crossover period, the PANAS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal total score means were calculated for the negative affect using a linear mixed model regression that controlled for baseline and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 19.93 (1.18) | 19.5 (1.47)
  Day 1 | 21.63 (1.18) | 19.5 (1.47)
  Day 2 | 19.67 (1.26) | 19.72 (1.47)
  Day 3 | 19.11 (1.26) | 20.83 (1.47)
  Day 7 | 20.33 (1.18) | 22.39 (1.47)
  Day 14 | 20.78 (1.26) | 20.94 (1.47)
  Day 21 | 21.22 (1.26) | 21.94 (1.47)

16. Secondary Outcome: Clinician-Administered Dissociative States Scale (CADSS) Mean Total Score
Description: The Clinician Administered Dissociative States Scale (CADSS) mean total score at 230 minutes and 1, 2, 3, 7, 14, and 21 days following the first treatment administration. The CADSS is a 28-item clinician-rated assessment of dissociative states in the moment and contains both subjective and objective items. Items are rated on a scale of 0 to 4 (0 = not at all, 4 = extreme) with total score range between 0 and 112. A higher score indicates more severe dissociation. For each crossover period, the CADSS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose. Estimated marginal CADSS total score means were calculated using a linear mixed model regression that controlled for baseline and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 1.24 (0.24) | 1.98 (0.65)
  Day 1 | 1.54 (0.24) | 1.76 (0.65)
  Day 2 | 1.05 (0.25) | 0.98 (0.65)
  Day 3 | 0.94 (0.25) | 1.2 (0.65)
  Day 7 | 0.84 (0.24) | 1.43 (0.65)
  Day 14 | 1.17 (0.25) | 0.31 (0.65)
  Day 21 | 1.39 (0.25) | 1.2 (0.65)

17. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Mean Total Score
Description: The Brief Psychiatric Rating Scale (BPRS) mean total score at 230 minutes, 1 and 21 days following the first treatment administration. The BPRS is an 18-item clinician-rated scale that evaluates symptoms and behaviors that are characteristic of schizophrenia (e.g., hallucinations, unusual thought content). Each item is rated on scale of 1 (symptom not reported or observed) to 7 (very severe), with a total score range between 18 to 126. Higher scores indicate more severe symptoms of psychosis. For each crossover period, the BPRS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1 and 21 days days following the first dose. Estimated marginal BPRS total score means were calculated using a linear mixed model regression that controlled for baseline and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, and 1 and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 30.28 (1.31) | 30.33 (1.2)
  Day 1 | 29.88 (1.31) | 30.44 (1.2)
  Day 21 | 30.93 (1.39) | 32.1 (1.2)

18. Secondary Outcome: The Young Mania Rating Scale (YMRS) Total Score
Description: The Young Mania Rating Scale (YMRS) mean total score at 230 minutes, 1 and 21 days following the first treatment administration. The YMRS is an 11-item clinician-rated scale that evaluates symptoms of mania or hypomania in adults. Each item is rated on scale from either 0-4 or 0-8, where 0 indicates a symptom is not present, and the highest score (4 or 8) indicates a symptom is extremely severe, with a total score range between 0 and 60. Higher scores indicate more severe manic/hypomanic symptoms. For each crossover period, the YMRS was completed 1440 minutes (24 hours) before intervention (baseline) and 230 minutes, 1 and 21 days following the first dose. Estimated marginal total score means were calculated using a linear mixed model regression that controlled for baseline and allowed treatment differences to vary by time point.
Time Frame: 230 minutes, 1, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Units on a scale
  230 minutes | 2.08 (0.72) | 1.77 (0.53)
  Day 1 | 2.88 (0.72) | 1.33 (0.53)
  Day 21 | 1.94 (0.76) | 1.66 (0.53)

19. Secondary Outcome: Number of Participants With Suicide Ideation Assessed Using the Columbia Suicide Severity Rating Scale (CSSRS)
Description: Number of participants with suicide ideation assessed using the Columbia Suicide Severity Rating Scale (CSSRS) ideation score. The CSSRS is administered as a structured clinical interview, and a participant's responses to screening items determine which subsequent items are administered. CSSRS ideation scores can range from 0 to 5. Due to skew, CSSRS total score was dichotomized so that score of 0 indicated no suicidal ideation and score ≥1 indicated the presence of suicidal ideation. For each crossover period, the CSSRS was completed one day before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Participants
  230 minutes | 2 | 2
  Day 1 | 2 | 2
  Day 2 | 3 | 1
  Day 3 | 2 | 1
  Day 7 | 2 | 2
  Day 14 | 2 | 3
  Day 21 | 1 | 2

20. Secondary Outcome: Number of Participants With Suicide Ideation Assessed Using the Scale for Suicidal Ideation (SSI)
Description: Number of participants with suicide ideation assessed using the Scale for Suicide Ideation (SSI). SSI measures current suicidal ideation and behavior administered as a structured clinical interview, and a participant's responses to screening items determine which subsequent items are asked. A participant is asked from 5 and up to 21 items with each item rated on the scale of 0 to 2. Total scores range between 0 to 42. Due to skew, SSI total score was dichotomized so that score ≤1 indicated no suicidal ideation and score ≥2 indicated the presence of suicidal ideation. For each crossover period, the SSI was completed one day before intervention (baseline) and 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose.
Time Frame: 230 minutes, 1, 2, 3, 7, 14, and 21 days following the first dose for each intervention period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TS-161 | Placebo
Number analyzed (Participants) | 10 | 9
Participants
  230 minutes | 2 | 3
  Day 1 | 2 | 4
  Day 2 | 2 | 3
  Day 3 | 3 | 4
  Day 7 | 3 | 3
  Day 14 | 3 | 4
  Day 21 | 3 | 4

ADVERSE EVENTS:
Time Frame: Up to 16 weeks from start of study
Arm/Group | TS-161 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 7/11 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TS-161 (N=11) | Placebo (N=9)
Chest pain (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Hiccups (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Energy increased (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Feeling of body temperature change (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rectal tenesmus (Musculoskeletal and connective tissue disorders) | 1 | 0
Abnormal dreams (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 1 | 2
Hypersomnia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1
Vertigo (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Derealisation (Psychiatric disorders) | 1 | 0
Distractibility (Psychiatric disorders) | 1 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0
Tinea pedis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT04821271/Prot_SAP_000.pdf